CLINICAL TRIAL: NCT03354611
Title: Contrast-Enhanced Cone Beam Breast CT for Diagnostic Breast Imaging
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study progress doesn't meet the sponsor's requirement
Sponsor: Koning Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-01
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects in this group will be enrolled from screening assigned BIRADS 0, patient complaint, or referral for second opinion. The enrolled patient will accept CE-CBBCT scans within 4 weeks of her diagnostic mammography and before breast biopsy if biopsy is needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic Workup (Experimental): The subjects will first have a pre-contrast CBBCT scan. Iodinated contrast will be injected intravenously, and then another CBBCT scans will be performed to capture the tumor vasculature enhancement.
  Interventions: Radiation: Contrast Enhanced Cone Beam Breast CT Scan; Drug: Contrast Dye, Iodinated

INTERVENTIONS:
Radiation: Contrast Enhanced Cone Beam Breast CT Scan — * Pre-contrast scan
  * Begin contrast injection (and saline chaser)
  * Post-contrast Scan. Start time of post-contrast CE-CBBCT scan is 90-200 seconds after start of injection, depending on method of contrast delivery (bolus vs hand injection)
Drug: Contrast Dye, Iodinated — 1.5-2ml/kg body weight (100 ml maximum) of a low osmolar, nonionic, 300-350 mgI/ml iodinated contrast agent, will be injected at a rate of ~2.0 ml/s, for a total injection time of 30-60 seconds (for a 50 kg subject). This will be immediately followed by a saline "chaser" from 20 to 40 ml at ~2 ml/s (20 seconds) to maximize dynamic enhancement.

SUMMARY:
Up to one hundred (100) female patients will be enrolled and consented to participate in the study. These women will be enrolled from screening assigned BIRADS 0, patient complaint, or referral for second opinion. The enrolled patient will accept CE-CBBCT scans within 4 weeks of her diagnostic mammography and before breast biopsy if biopsy is needed. The final diagnostic workup outcome of these enrolled patients needs to include at least 30 confirmed cancers cases.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 35 years or older
* Any ethnicity
* Have an abnormality detected by Breast Self Exam (BSE), or Clinical Breast Exam (CBE), or have an abnormality detected by an imaging modality.
* Will undergo study imaging within four weeks from the date of diagnostic mammography, prior to breast biopsy (if needed).
* Able to provide informed consent
* Post-menopausal, surgically sterile, or effective birth control. For women of childbearing potential, negative pregnancy test or has signed pregnancy test waiver
* If required by standard of care, eGFR >45 within 48 hours to 6 weeks of CE-CBBCT exam

Exclusion Criteria:

* Pregnancy
* Lactation
* Unknown pregnancy status AND
* has refused pregnancy testing and
* has refused to sign a pregnancy test waiver
* Women who are unable or unwilling to understand or to provide informed consent
* Women with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Women who are unable to tolerate study constraints.
* Women who have received radiation treatments to the thorax or breast area for malignant and nonmalignant conditions, such as (but not limited to):

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkin's disease
  * Women who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
  * Women who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to):
* Tuberculosis
* Severe scoliosis

Additional Exclusion Criteria Due To Contrast Injection:

* Allergic to iodinated contrast material
* Previous non-ionic contrast reaction
* Any conditions below regardless of eGFR

  * Renal Disease
  * Chronic renal dysfunction
  * Renal Transplant (or waiting for a transplant)
  * One kidney or other birth defect
  * Polycystic Kidneys
  * Renal Tumor/Renal Cancer
  * History of liver failure/cirrhosis/liver transplant/pending liver transplant
  * Congestive heart failure
  * Multiple myeloma
  * Hyperthyroidism
  * Pheochromocytoma
  * Sickle Cell Disease
  * Asthma requiring daily use of inhaler Additional exclusion criteria due to machine limitations
* Patient's body weight is over the limit of the scanner table (440 lbs or 200kg)

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Breast lesions | Within 4 weeks after the imaging acquisition if finished if there is a suspicious finding in the images.
  The existence of lesions in the breast

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UR Medicine Breast Imaging, Rochester, New York
  - Knoxville Comprehensive Breast Center, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connell A, Conover DL, Zhang Y, Seifert P, Logan-Young W, Lin CF, Sahler L, Ning R. Cone-beam CT for breast imaging: Radiation dose, breast coverage, and image quality. AJR Am J Roentgenol. 2010 Aug;195(2):496-509. doi: 10.2214/AJR.08.1017. PMID 20651210
- [Background] Pediconi F, Venditti F, Padula S, Roselli A, Moriconi E, Giacomelli L, Catalano C, Passariello R. CE-Magnetic Resonance Mammography for the evaluation of the contralateral breast in patients with diagnosed breast cancer. Radiol Med. 2005 Jul-Aug;110(1-2):61-8. English, Italian. PMID 16163140
- [Background] Esserman L, Hylton N, Yassa L, Barclay J, Frankel S, Sickles E. Utility of magnetic resonance imaging in the management of breast cancer: evidence for improved preoperative staging. J Clin Oncol. 1999 Jan;17(1):110-9. doi: 10.1200/JCO.1999.17.1.110. PMID 10458224
- [Background] Orel SG, Schnall MD. MR imaging of the breast for the detection, diagnosis, and staging of breast cancer. Radiology. 2001 Jul;220(1):13-30. doi: 10.1148/radiology.220.1.r01jl3113. PMID 11425968
- [Background] Gulsun M, Demirkazik FB, Ariyurek M. Evaluation of breast microcalcifications according to Breast Imaging Reporting and Data System criteria and Le Gal's classification. Eur J Radiol. 2003 Sep;47(3):227-31. doi: 10.1016/s0720-048x(02)00181-x. PMID 12927667
- [Background] McDonald RJ, McDonald JS, Kallmes DF, Jentoft ME, Murray DL, Thielen KR, Williamson EE, Eckel LJ. Intracranial Gadolinium Deposition after Contrast-enhanced MR Imaging. Radiology. 2015 Jun;275(3):772-82. doi: 10.1148/radiol.15150025. Epub 2015 Mar 5. PMID 25742194
- [Background] Prionas ND, Lindfors KK, Ray S, Huang SY, Beckett LA, Monsky WL, Boone JM. Contrast-enhanced dedicated breast CT: initial clinical experience. Radiology. 2010 Sep;256(3):714-23. doi: 10.1148/radiol.10092311. PMID 20720067
- [Background] Seifert P, Conover D, Zhang Y, Morgan R, Arieno A, Destounis S, Somerville P, Murphy PF. Evaluation of malignant breast lesions in the diagnostic setting with cone beam breast computed tomography (Breast CT): feasibility study. Breast J. 2014 Jul-Aug;20(4):364-74. doi: 10.1111/tbj.12285. Epub 2014 Jun 17. PMID 24934253
- [Background] O'Connell AM, Kawakyu-O'Connor D. Dedicated Cone-beam Breast Computed Tomography and Diagnostic Mammography: Comparison of Radiation Dose, Patient Comfort, And Qualitative Review of Imaging Findings in BI-RADS 4 and 5 Lesions. J Clin Imaging Sci. 2012;2:7. doi: 10.4103/2156-7514.93274. Epub 2012 Feb 25. PMID 22439131
- [Background] O'Connell AM, Karellas A, Vedantham S. The potential role of dedicated 3D breast CT as a diagnostic tool: review and early clinical examples. Breast J. 2014 Nov-Dec;20(6):592-605. doi: 10.1111/tbj.12327. Epub 2014 Sep 8. PMID 25199995
- [Background] Fukumura D, Duda DG, Munn LL, Jain RK. Tumor microvasculature and microenvironment: novel insights through intravital imaging in pre-clinical models. Microcirculation. 2010 Apr;17(3):206-25. doi: 10.1111/j.1549-8719.2010.00029.x. PMID 20374484
- [Background] Boetes C, Mus RD, Holland R, Barentsz JO, Strijk SP, Wobbes T, Hendriks JH, Ruys SH. Breast tumors: comparative accuracy of MR imaging relative to mammography and US for demonstrating extent. Radiology. 1995 Dec;197(3):743-7. doi: 10.1148/radiology.197.3.7480749.

DOCUMENTS (1):
  • Study Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03354611/Prot_002.pdf